CLINICAL TRIAL: NCT05010629
Title: Phase 2 Study of 9-ING-41, a Glycogen Synthase Kinase 3 Beta (GSK 3β) Inhibitor, Plus Carboplatin in Patients With Advanced, Metastatic Salivary Gland Carcinoma
Brief Title: 9-ING-41 Plus Carboplatin in Salivary Gland Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn J. Hanna (Other)
Collaborators: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, Glenn J. Hanna, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-384
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Salivary Gland Cancer; Recurrent Salivary Gland Cancer; Metastatic Cancer; Adenoid Cystic Carcinoma
Keywords: Salivary Gland Cancer; Recurrent Salivary Gland Cancer; Metastatic Salivary Gland Cancer; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Neoplasm Metastasis; Carcinoma, Adenoid Cystic | interventions — 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 9-ING-41 + carboplatin (Experimental): Participants will be divided into 2 cohorts: Salivary Gland Cancer with adenoid cystic carcinoma (ACC) and Salivary Gland Cancer without adenoid cystic carcinoma (ACC) and receive:
  * 9-ING-41 2x every 21 day study cycle on Day 1 and Day 4 up to 1 year with option to continue beyond if participant is showing benefit
  * Carboplatin 1x every 21 day study cycle on Day 1 up to 1 year
  Interventions: Drug: 9-ING-41; Drug: Carboplatin

INTERVENTIONS:
Drug: 9-ING-41 — Intravenous infusion
Drug: Carboplatin — Intravenous infusion
  Other Names: Paraplatin

SUMMARY:
This trial is investigating an intravenous (IV) medication called 9-ING-41 in combination with chemotherapy (carboplatin) for the treatment of advanced salivary gland cancers.

The names of the study drug(s) involved in this study are:

* 9-ING-41 (a GSK-3β inhibitor)
* Carboplatin chemotherapy

DETAILED DESCRIPTION:
This is a phase 2, open-label, non-randomized, single institution study investigating the novel glycogen synthase kinase-3 beta (GSK-3β) inhibitor 9-ING-41 in combination with carboplatin chemotherapy in patients with incurable, recurrent or metastatic salivary gland carcinomas (SGC).

The U.S. Food and Drug Administration (FDA) has not approved 9-ING-41 as a treatment for any disease. Carboplatin is used as a treatment for salivary gland cancers, and is approved by the FDA for many cancer types.

9-ING-41 has been identified in other studies as a therapy to block the over-expression of the glycogen synthase kinase-3 beta (GSK-3β) protein, which is thought to be important in signaling cancer growth and to have immune properties. It is believed that GSK-3β is over-expressed in salivary gland cancers and by blocking the action of GSK-3β protein with 9-ING-41 it could slow salivary cancer cell growth that have developed resistance to prior chemotherapy exposure.

The research study procedures include screening for eligibility and study treatment including evaluations and follow-up visits roughly every 3-weeks while on therapy, for up to one year as long as disease does not get worse and the drug therapy remains safe and tolerable.

It is expected that about 33 people treated will take part in this research study.

Actuate Therapeutics is supporting this research study by providing the study drug (9-ING-41) and funding some of the logistics of the trial that are beyond what would be considered standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed salivary gland carcinoma (any histologic subtype, including ACC) with evidence of recurrent, metastatic or advanced, unresectable disease.
* Willing to provide tumor tissue from a diagnostic biopsy or prior surgery.
* Age 18 years or older
* ECOG performance status 0-2 (see Appendix A)
* Participant must have organ and marrow function as defined below within 14 days prior to study registration:

  * leukocytes ≥ 3,000/mcL
  * absolute neutrophil count ≥ 500/mcL
  * hemoglobin ≥ 8.5 g/dL
  * platelets ≥ 75,000/mcL
  * total bilirubin ≤ 2.0 g/dL
  * AST(SGOT)/ALT(SGPT) ≤ 2.5× institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥50 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Participants must have documentation of a new or progressive lesion on a radiologic imaging study performed within 12 months prior to study registration (progression of disease over any interval is allowed) and/or new or worsening disease-related symptoms within 12 months prior to study registration. This assessment is performed by the treating investigator. Evidence of progression by RECIST v1.1 criteria not required.
* Participants must have at least one RECIST v1.1 measurable non-CNS based lesion, as defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) ≥ 1 cm with CT scans or MR imaging.
* Prior systemic therapy: At least 2 weeks must have elapsed since the end of prior chemotherapy, biological agents (3 weeks for anti-cancer monoclonal antibody containing regimens) or any investigational drug product, with adequate recovery of treatment-related toxicity to NCI CTCAE Version 5.0 grade ≤1 (or tolerable grade 2) or back to baseline (except for alopecia or neuropathy). Any number of prior therapies for recurrent/metastatic SGC are permitted (including prior carboplatin exposure); but prior therapy for recurrent/metastatic SGC is not required for participation.
* Ability to understand and the willingness to sign a written informed consent document.

Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days of study registration. Female subjects of childbearing potential should have a negative urine or serum pregnancy test repeated within 72 hours prior to receiving the first dose of study medication. WOCBP will be instructed to adhere to contraception for a period of 90 days after the last dose of investigational product. "Women of childbearing potential (WOCBP)" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level greater than 40 mIU/mL.

* Men who are sexually active with WOCBP must agree to use any contraceptive method with a failure rate of less than 1% per year. Men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 90 days after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception. See Appendix B for further guidance on contraception.

Exclusion Criteria:

* Metastatic disease impinging on the spinal cord or threatening spinal cord compression. Patients that have had previous treatment of disease with impinging on the cord with either surgery or radiotherapy with clinical or radiographic evidence of response or stability are eligible.
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment), and have no evidence of new or enlarging brain metastases.
* Concurrent administration of other cancer specific therapy or investigational agents during the course of this study is not allowed.
* Patients on anticoagulants that require INR monitoring (such as warfarin).
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant or lactating women.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include: basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and low-risk prostate adenocarcinoma being managed with active surveillance. A history of another separate malignancy in remission without evidence of active disease in the last 2 ears is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Best Overall response rate | Up to 1 year
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Measured with RECIST v 1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 1 year
  Progression-Free Survival (PFS) is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Overall Survival (OS) | Up to 2 years
  Overall Survival (OS) is defined as the time from study registration to death due to any cause, or censored at date last known alive
Duration of therapeutic response | Up to 2 years
  Assessed using RECIST v1.1
Duration of therapeutic response Cohort 1 | Up to 2 years
  Assessed using RECIST v1.1
Duration of therapeutic response Cohort 2 | Up to 2 years
  Assessed using RECIST v1.1
Number of Participants with treatment related Adverse Events per CTCAE 5.0 | Up to 2 years
  Assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
University of Washington Quality of Life Questionnaire (UW-QOL) Response | Baseline, 12 weeks up to 1 year
  Descriptive statistics from the questionnaire will be summarized across timepoints of assessment. Rates of drop-out/non-response to QOL assessments and corresponding reason will also be summarized across timepoints of assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Hanna, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu